CLINICAL TRIAL: NCT02959515
Title: The Effects of Different Methods of Non-ventilated Lung Management on Oxygen Delivery (DO2) During One Lung Ventilation (OLV) in the Supine Position for Video Assisted Thoracoscopic (VATS) Atrial Fibrillation Ablation
Brief Title: The Effects of Different Types of Non-ventilated Lung Management on DO2 During OLV in the Supine Position
Acronym: OLVinFACHIR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro Cardiologico Monzino (Other)
Responsible Party: Principal Investigator, luca salvi, Anesthesia & ICU Senior consultant, Centro Cardiologico Monzino
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CentroCM
Record Dates: First submitted 2016-10-26; First posted 2016-11-09 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-10

CONDITIONS: One-Lung Ventilation; Thoracic Surgery Video Assisted; Supine Position
MeSH Terms: conditions — Deception

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Capnothorax (Active Comparator): Capnothorax is obtained by the insufflation of CO2in the right pleural cavity and maintained at a preset pressure of 10 mmHg .Arterial and central venous blood gasanalyses, hemodynamic and respiratory variables will be recorded.
  Interventions: Procedure: Capnothorax
- Capnothorax and CPAP (Active Comparator): Capnothorax is obtained by the insufflation of CO2in the right pleural cavity and maintained at a preset pressure of 10 mmHg. CPAP on the non ventilated lung is set at 10 cm H2O and FiO2=1. Arterial and central venous blood gasanalyses, hemodynamic and respiratory variables will be recorded.
  Interventions: Procedure: Capnothorax and CPAP

INTERVENTIONS:
Procedure: Capnothorax — Insufflation of CO2 at a preset pressure of 10 cmH2O in the right pleural cavity.
  Arms: Capnothorax
Procedure: Capnothorax and CPAP — Insufflation of CO2 at a preset pressure of 10 cmH2O in the right pleural cavity.
  Continuous positive airway pressure of 10 cmH2O delivered by CF 800 Continuous flow CPAP, Drager.
  Arms: Capnothorax and CPAP

SUMMARY:
The aim of this study is the comparison of oxygen delivery during OLV+capnothorax and OLV+capnothorax and CPAP.

DETAILED DESCRIPTION:
One-lung ventilation (OLV) is utilized mainly during thoracic procedures when surgeon needs the lung deflated to expose the surgical field. In this situation both lungs are perfused but only one is ventilated resulting in high grade of shunt and eventually hypoxemia .

Most of thoracic procedures are performed with the pt lying on one side; the deflated lung receive less blood flow both for the gravity and for the hypoxic pulmonary vasoconstriction (HPV) thus reducing the shunt.

If the pt lyes supine, as in VATS atrial fibrillation (AF) surgical ablation, the protective effect of gravity is lost, shunt remains high and severe hypoxemia is common. Some algorithms are used to improve oxygenation during OLV: high fraction of inspired oxygen (FiO2), positive end expiratory pressure (PEEP) on the ventilated lung, continuous positive airway pressure (CPAP) on the deflated lung, but the latter can be used with caution during VATS because of the obstruction of the surgical field. Increasing the pressure in the pleural cavity with carbon dioxyde (CO2) (capnothorax) could decrease the blood flow in the deflated lung, helping in reducing shunt but this is not yet demonstrated and this manouver could decrease cardiac output. The oxygen delivery (DO2) is cardiac output (CO) by oxygen content and during this surgery both these factors could be compromised.

All consecutive pts electively subjected to OLV in supine position for VATS ablation of AF will be enrolled. On the day of surgery pts will be randomly allocated in two groups depending on the management of the non-ventilated lung (capnothorax or capnothorax and CPAP.

Pts in supine position; tracheal intubation with left-sided double lumen tube (DLT) and position confirmed by bronchoscopy. Lungs are initially ventilated with pressure controlled mode (PCV) at a tidal volume (TV) of 7 mL/kg, I:E ratio 1:2, respiratory rate (RR) to obtain a PaCO2 40-45 mmHg, FiO2 =1 and PEEP 5 cm H2O. During OLV inspiratory pressure is reduced to obtain a TV of 5 mL/Kg, maintaining FiO2=1, PEEP 5 cm H2O and adjusting RR to obtain a PaCO2 40-45 mmHg. Capnothorax is obtained by the insufflation of CO2 and maintained at a preset pressure of 10 mmHg. CPAP on the non ventilated lung is set at 10 cm H2O and FiO2=1.

After institution of OLV pts will be randomized to receive capnothorax alone (Group CA) or to receive capnothorax and CPAP (Group CC)

Arterial and central venous blood gasanalyses, hemodynamic and respiratory variables will be recorded at the following points:

a) spontaneous breathing at FiO2=0.21; b) 10' after double lung ventilation (TLV); c) 10'after OLV; d) 10' after OLV and capnothorax (Group CA) or OLV, capnothorax and CPAP (Group CC) e) double lung ventilation (TLV) at the end of the surgical procedure Differences of DO2, shunt fraction (QS/QT), and derived variables between the two groups will be tested by T-test.

40 pts (20 per groups) will allow 80% power to deem as significant (alpha = 0.05) a difference of 50 mL/min in DO2 (with standard deviation of 50 mL/min) between the two managements of the non-ventilated lung.

If SaO2 will decrease below 90% an alveolar recruitment strategy will be performed and if not effective TLV will be initiated together with dropping the pt out of the study

ELIGIBILITY:
Inclusion Criteria:

* Pts electively subjected to OLV in supine position for VATS ablation of AF and requiring OLV for > 30'

Exclusion Criteria:

* Expected difficult positioning of DLT, severe obesity BMI > 35, uncompensated cardiac disease. OLV < 30'.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-03 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Oxygen delivery | 10 min after institution of capnothotax or capnothorax and CPAP
  Oxygen delivery is cardiac output times arterial oxygen content

SECONDARY OUTCOMES:
Pulmonary shunt | 10 min after institution of capnothotax or capnothorax and CPAP
  Fraction of venous blood which is not oxygenated by the lungs

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Cardiologico Monzino, Milan, Italy